CLINICAL TRIAL: NCT03544918
Title: Prevalence of Congenital Long QT Syndrome and Acquired QT Prolongation in a Hospital Cohort
Status: Completed | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jan Hysing MD PhD, MD PhD cardiologist consultant, Sykehuset Telemark
Other Study IDs: REK 2013/1090
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples for DNA Analysis. Parafin embeded tissue will be used as well
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with long QT syndrome.: Patents with Long QT syndrome hospitilized. To be followed over time with no intervention. Observational study.
- Patients in Telemark with normal QT time: Patients in Telemark with normal QT time. To be followed over time with no intervention. Observational study.

SUMMARY:
The Long QT syndrome is associated with potentially life-threatening cardiac arrhythmias as ventricular tachycardia (Torsade de pointes) as well as ventricular fibrillation, and might lead to syncope as well as sudden cardiac death (1). Good results have been achieved by treating patient at risk with beta blockers and implantable cardiac defibrillator (ICD). It is therefore important to diagnose the condition as early as possible as the disease is treatable (2).

Prolonged QT duration might also be induced by the intake of numerous pharmaceutical substances, as well as with electrolyte disturbances, which also increases the risk of life-threatening cardiac arrhythmias. Furthermore, congenital LQTS can arise from mutations in one of at least 13 different genes. Many of these genes encode proteins which are constituents of ion channels. The genetically defined long QT syndrome has autosomal dominant (Romano Ward Syndrome) or autosomal recessive (Jervell and Lange-Nielsen Syndrome) inheritance.

In this study we are using the hospital ECG database obtained with the GE Marquette 12SL ECG Analysis Program® at Telemark Hospital Skien recorded between March 2004 and April 2014. This database stores approximately 200 000 ECG recordings from 60 000 unique patients.

By using the search algorithm in the MUSE ECG database, 2398 recordings have been be identified from 1603 patients where the corrected QT time is longer than 500 ms, and QRS is less than 120 ms.

ECG recordings with QT intervals longer than 500 ms represents less than 1% of the population (5). Individuals having these recordings are selected for extensive clinical follow up. The patients will be offered the opportunity to have genetic analysis performed in order to distinguish between inherited or acquired long QT syndrome. The appropriate treatment will be initiated according to guidelines for patients with inherited QT syndrome. For patients with aquired long QT syndrome substitution of unfavourable pharmacotherapy or correction of electrolytes shall be performed in order to reduce their risk of cardiac arrhythmias.

A T wave morphology score gives independent prognostic information useful for risk stratification. The purpose of this substudy is to examine if the T wave morphology score applied on the 1531 patients ECGs with QTc >500 ms, has independent prognostic value in this cohort.

DETAILED DESCRIPTION:
2. PURPOSE OF THE STUDY

The study has the intention to:

* Identify patients with inherited LQTS in order to give them optimal treatment.
* To identify patients with acquired QT prolongation in order to possibly correct electrolyte disorders and therapeutically prescriptions in order to minimize the chance of life-threatening arrhythmias.
* To analyse to what extend a specific reason for QT prolongation can be found in patients with heart rate adjusted QT prolongation, or to which extend the QT prolongation without syncope, or family history of sudden cardiac death, is an unspecific finding.
* To analyse time dependent risk of patients with QT prolongation related to underlying disease
* To analyse to what extend genetic variations might predispose for acquired QT prolongation.
* To compare life expectancy of patients with QT prolongation related to case control patients with out QT prolongation.
* To implement rapid reaction on newly diagnosed QT prolongation, and follow up of survival after implementation of improved care.

  * To examine if the T wave morphology score applied on patients ECGs with QTc >500 ms, has independent prognostic value in this cohort.

ELIGIBILITY:
Inclusion Criteria:

QT time in EKG more Tham 500 ms -

Exclusion Criteria:

Patient refuses to be a part of the study registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Long QT syndrome is associated with potentially life-threatening cardiac arrhythmias.
  In this study we are using the hospital ECG database obtained with the GE Marquette 12SL ECG Analysis Program® This database stores approximately 200 000 ECG recordings from 60 000 unique patients.
  By using the search algorithm in the MUSE ECG database, 2398 recordings have been be identified from 1603 patients where the corrected QT time is longer than 500 ms, and QRS is less than 120 ms.
Sampling Method: Non-Probability Sample
Enrollment: 1536 (Actual)
Dates: Start 2015-06; Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
survival | 2004-2014
  Death certificate information from national register

SECONDARY OUTCOMES:
comorbidity data from hospital database Genetic defects data | 2004-2014
  Data extracted from hospital notes

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hysing, PhD, Principal Investigator — Sykehuset Telemark
Locations (1):
- Sykehuset Telemark, Skien, Telemark, Norway

IPD SHARING:
Plan to Share IPD: Undecided